CLINICAL TRIAL: NCT04243304
Title: Longitudinal Measurement of Synaptic Density to Monitor Progression of Parkinson's Disease.
Brief Title: Synaptic Density and Progression of Parkinson's Disease.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: s61477
Record Dates: First submitted 2020-01-10; First posted 2020-01-28 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; PET; UCB-J; PE2I
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Longitudinal study design (2 years follow up) where results of SV2A PET/CT, PE2I PET/MR and clinical rating scales are compared between PD patients and healthy controls.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PD patients (Experimental): At baseline and 2-year follow-up
  Interventions: Other: 11C-UCB-J PET-CT; Other: 18F-PE2I PET-MR
- Healthy controls (Active Comparator): At baseline and 2-year follow-up
  Interventions: Other: 11C-UCB-J PET-CT; Other: 18F-PE2I PET-MR

INTERVENTIONS:
Other: 11C-UCB-J PET-CT — Positron Emission Tomography (PET) of synaptic vesicle protein 2A (SV2A) using the radioligand 11C-UCB-J.
Other: 18F-PE2I PET-MR — Positron Emission Tomography (PET) of dopamine transporter (DAT) using the radioligand 18F-FE-PE2I, and brain MRI performed simultaneously.

SUMMARY:
AIM: To assess synaptic density and to investigate the potential relationship of regional synaptic loss with motor and non-motor symptoms and with disease progression in the human brain in vivo in patients with PD.

DESIGN: We will include 30 PD patients and 20 healthy controls. All subjects will undergo a clinical examination, with comprehensive assessment of motor and non-motor symptoms, and imaging evaluation consisting of 11C-UCB-J PET-CT and 18F-FE-PE2I PET-MR at baseline and after 2 years.

ELIGIBILITY:
Inclusion Criteria:

* PD diagnosis based on MDS clinical diagnostic criteria for Parkinson's disease
* Less than 5 years disease duration since motor symptom onset according to the patient
* Hoehn-Yahr stage 1 or 2 in medication ON state
* Capacity to understand the informed consent form

Exclusion Criteria:

* Neuropsychiatric diseases other than PD
* Major internal medical diseases
* Relevant abnormalities on MR brain
* History of alcohol or drug abuse
* Contraindications for MR
* Pregnancy
* Previous participation in other research studies involving ionizing radiation with > 1 mSv over past 12 months.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Baseline differences in synaptic density. | Data analysis wel be done when all subjects have undergone the baseline evaluation.
  Baseline differences (%) in synaptic density between patients and controls.
Correlations between clinical scores and synaptic density. | Data analysis wel be done when all subjects have undergone the 2-year follow-up evaluation.
  Correlations between clinical scores and synaptic density in the patient group.
Differences in the rate of decline of synaptic density. | Data analysis wel be done when all subjects have undergone the 2-year follow-up evaluation.
  Differences (%) in the rate of decline of synaptic density between patients and controls.
Correlations between progression of the clinical scores and decline of synaptic density. | Data analysis wel be done when all subjects have undergone the 2-year follow-up evaluation.
  Correlations between progression of the clinical scores and decline of synaptic density in the patient group.

SECONDARY OUTCOMES:
Baseline differences in DAT levels. | Data analysis wel be done when all subjects have undergone the baseline evaluation.
  Baseline differences (%) in DAT levels between patients and controls.
Correlations between clinical scores and DAT levels. | Data analysis wel be done when all subjects have undergone the 2-year follow-up evaluation.
  Correlations between clinical scores and DAT levels in the patient group.
Differences in the rate of decline of global and DAT levels. | Data analysis wel be done when all subjects have undergone the 2-year follow-up evaluation.
  Differences (%) in the rate of decline of global and DAT levels between patients and controls.
Correlations between progression of the clinical scores and decline of DAT levels. | Data analysis wel be done when all subjects have undergone the 2-year follow-up evaluation.
  Correlations between progression of the clinical scores and decline of DAT levels in the patient group.

CONTACTS AND LOCATIONS:
Overall Officials: Wim Vandenberghe, MD, PhD, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Needs to be decided.